CLINICAL TRIAL: NCT00005596
Title: ALinC 17: Protocol for Patients With Newly Diagnosed Standard Risk Acute Lymphoblastic Leukemia (ALL): A Phase III Study
Brief Title: Combination Chemotherapy in Treating Children With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9905; COG-P9905 (Other: Children's Oncology Group); POG-9905 (Other: Pediatric Oncology Group); CDR0000067704 (Other: Clinical Trials.gov); NCI-2012-02325 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Leucovorin; Mercaptopurine; Methotrexate; pegaspargase; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive IT methotrexate on day 1 followed by methotrexate IV over 20 minutes followed by methotrexate continuously over 23.6 hrs on wks 7, 10, 13, 16,19, and 22. At 42 hrs after the beginning of the methotrexate infusion, patients receive oral leucovorin calcium every 6 hrs for a total of 3 doses. Patients also receive oral mercaptopurine daily beginning on wk 5 and continuing until the completion of consolidation therapy; oral dexamethasone twice daily on days 1-7 of wks 8 and 17; and vincristine sulfate IV on day 1 of wks 8, 9, 17, and 18.
  Interventions: Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate
- Arm II (Experimental): Patients receive methotrexate IV over 4 hours on weeks 7, 10, 13, 16, 19, and 22. At 42 hours after the beginning of the methotrexate infusion, patients receive oral leucovorin calcium as in arm I. Patients also receive mercaptopurine, dexamethasone, vincristine sulfate, and IT methotrexate as in arm I.
  Interventions: Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate
- Arm III (Experimental): Patients receive methotrexate IV as in arm I on weeks 7, 10, 13, 24, 27, and 30; leucovorin calcium as in arm I; pegaspargase IM on day 2, 3, OR 4 of wk 16; oral mercaptopurine daily on wks 5-13, and from wk 24 until the completion of consolidation therapy. Patients also receive IT methotrexate as in arm I on wks 7, 10, 13, 16, 20, 21, and 30; oral dexamethasone 2x daily on weeks 8, 16-18, and 28 for a total of 35 days; vincristine sulfate IV on day 1 of wks 8, 9, 16, 17, 18, 28, and 29; daunorubicin hydrochloride IV on day 1 of wks 16-18; cyclophosphamide IV over 30 minutes on day 1 of week 20; cytarabine IV or subcutaneously daily on days 2-5 of wks 20 and 21; and oral thioguanine daily on wks 20-21.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate
- Arm IV (Experimental): Patients receive methotrexate IV as in arm II on weeks 7, 10, 13, 24, 27, and 30; leucovorin calcium as in arm I; and pegaspargase, mercaptopurine, IT methotrexate, dexamethasone, vincristine sulfate, daunorubicin hydrochloride, cyclophosphamide, cytarabine, and thioguanine as in arm III.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate

INTERVENTIONS:
Drug: cyclophosphamide
  Arms: Arm III; Arm IV
Drug: cytarabine
  Arms: Arm III; Arm IV
Drug: daunorubicin hydrochloride — 30 mg/m2 IV Day 1 of weeks 16, 17, and 18. Give Week 16 dose if ANC ≥ 500/μL and platelets ≥ 75,000/μL. Continue to give during Weeks 17 and 18, even in the face of uncomplicated myelosuppression
  Other Names: daunomycin
  Arms: Arm III; Arm IV
Drug: dexamethasone — 6 mg/m2/day divided BID for 7 days during weeks 8 and 17.
  Other Names: DEX
Drug: leucovorin calcium — 5 mg/m2/dose of leucovorin will be given PO q12h x 2 doses beginning 48 hours after the start of the MTX.
Drug: mercaptopurine — 50 mg/m2 dose po qhs Weeks 5 through 13 (total 9 wks) and from Week 24 until the end of consolidation. Only hold for uncomplicated myelosuppression, only if IV MTX course is delayed, until ANC > 500/μL and platelets > 75,000/uL
  Other Names: 6-MP
Drug: methotrexate — IV: 1 gm/m2 given as a 200 mg/m2 bolus over 20 min followed by 800 mg/m2 over 23.6 hours given during Weeks 7, 10, 13, 16, 19, and 22.
  IT: Doses by age, Weeks 7, 10, 13, 16, 19 and 22.
  Other Names: MTX
Drug: pegaspargase — 2,500 IU/m2 will be given IM x 1 on Days 2,3,or 4 of Week 16; > or = 1 day after the IT MTX
  Other Names: PEG
  Arms: Arm III; Arm IV
Drug: thioguanine — 60 mg/m2 po qhs during Weeks 20 and 21 (total 14 days). Start week 20 when ANC > or = 500/ul and platelets > or = 75,000/uL. Continue to give all 14 doses despite uncomplicated myelosuppression.
  Other Names: 6-TG
  Arms: Arm III; Arm IV
Drug: vincristine sulfate — 1.5 mg/m2 IV on Day 1 of Weeks 8, 9, 17 and 18 (max 2 mg)
  Other Names: VCR

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which regimen of chemotherapy is more effective for acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is comparing four regimens of combination chemotherapy to see how well they work in treating children with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if multidrug delayed-intensification therapy improves outcome in children with newly diagnosed standard-risk acute lymphocytic leukemia.
* Compare the efficacy and toxicity of methotrexate administered over 4 hours vs methotrexate administered over 24 hours in this patient population.
* Determine the correlation between event-free survival, minimal residual disease, and early response in this patient population treated with this multiple drug regimen.

OUTLINE: This is a randomized, multicenter study.

* Induction (weeks 1-4): Patients receive induction therapy on POG 9900.
* Consolidation (weeks 5-32): Patients are randomized to one of four treatment arms. Patients with t(1;19) are randomized to either arm III or arm IV.

  * Arm I (weeks 5-24): Patients receive IT methotrexate (MTX) on day 1 followed by MTX IV over 20 minutes followed by MTX continuously over 23.6 hours on weeks 7, 10, 13, 16,19, and 22. At 42 hours after the beginning of the MTX infusion, patients receive oral leucovorin calcium every 6 hours for a total of 3 doses. Patients also receive oral mercaptopurine daily beginning on week 5 and continuing until the completion of consolidation therapy; oral dexamethasone twice daily on days 1-7 of weeks 8 and 17; and vincristine IV on day 1 of weeks 8, 9, 17, and 18.
  * Arm II (weeks 5-24): Patients receive MTX IV over 4 hours on weeks 7, 10, 13, 16, 19, and 22. At 42 hours after the beginning of the MTX infusion, patients receive oral leucovorin calcium as in arm I. Patients also receive mercaptopurine, dexamethasone, vincristine, and IT MTX as in arm I.
  * Arm III (weeks 5-32): Patients receive MTX IV as in arm I on weeks 7, 10, 13, 24, 27, and 30; leucovorin calcium as in arm I; pegaspargase IM on day 2, 3, OR 4 of week 16; and oral mercaptopurine daily on weeks 5-13, and from week 24 until the completion of consolidation therapy. Patients also receive IT MTX as in arm I on weeks 7, 10, 13, 16, 20, 21, and 30; oral dexamethasone twice daily on weeks 8, 16-18, and 28 for a total of 35 days; vincristine IV on day 1 of weeks 8, 9, 16, 17, 18, 28, and 29; daunorubicin IV on day 1 of weeks 16-18; cyclophosphamide IV over 30 minutes on day 1 of week 20; cytarabine IV or subcutaneously daily on days 2-5 of weeks 20 and 21; and oral thioguanine daily on weeks 20-21.
  * Arm IV (weeks 5-32): Patients receive MTX IV as in arm II on weeks 7, 10, 13, 24, 27, and 30; leucovorin calcium as in arm I; and pegaspargase, mercaptopurine, IT MTX, dexamethasone, vincristine, daunorubicin, cyclophosphamide, cytarabine, and thioguanine as in arm III.
* Intensive continuation (weeks 25-80): At weeks 25-72 for arms I and II, and at weeks 33-80 for arms III and IV, patients receive oral MTX every 6 hours for 4 doses on weeks 1, 3, 5, 7, 9, and 11; oral mercaptopurine daily; oral leucovorin calcium every 12 hours for 2 doses beginning 48 hours after the start of MTX; IT MTX and vincristine IV on day 1 of week 12; and oral dexamethasone twice daily on days 1-7, beginning with the administration of vincristine. Treatment repeats every 12 weeks for 4 courses.
* Additional continuation (weeks 73-130): At weeks 73-130 for arms I and II, and at weeks 81-130 for arms III and IV, patients receive oral MTX weekly; oral mercaptopurine daily; vincristine IV on day 1 every 12 weeks; oral dexamethasone as during intensive continuation therapy; and IT MTX on day 1 every 12 weeks, beginning with the last week of the first course (in place of oral MTX).

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then every 6-12 months for 1 year.

PROJECTED ACCRUAL: A total of 1,014 patients will be accrued for this study within 3.22 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of newly diagnosed B-precursor acute lymphocytic leukemia
* Standard risk (not low, high, or very high risk)
* Prior registration and treatment on POG 9900 Classification Study

PATIENT CHARACTERISTICS:

Age:

* 1 to 21 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1076 (Actual)
Dates: Start 2000-04; Primary Completion 2005-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Improvement in outcome in children receiving multidrug delayed-intensification therapy | Up to 4 years
  The overall plan is to accrue for 3.1 years or until all accrual goals have been met, whichever occurs first. Since power is determined by event-rates, lower or higher than expected event rates could lead to an amendment to alter the accrual goal. This consideration will be made independent of arm-specific outcome, in order to eliminate bias

SECONDARY OUTCOMES:
Event-free survival, minimal residual disease, and early response | 5 years
  The test statistic will compare Kaplan-Meier curves. Cox multiple regression will be utilized.
Occurrence of anticipated failures | Up to 5 years
  An O'Brien-Fleming analysis will be conducted.
Total grade 3+ central nervous system (CNS) toxicity rates based on the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naomi J. Winick, MD, Study Chair — Simmons Cancer Center
Locations (123):
- United States (108):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Stanford Cancer Center at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - University of Missouri - Columbia, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Beth Israel Medical Center - Singer Division, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
- University Medical Center Groningen, Groningen, Netherlands
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Background] Chen IM, Harvey RC, Mullighan CG, Gastier-Foster J, Wharton W, Kang H, Borowitz MJ, Camitta BM, Carroll AJ, Devidas M, Pullen DJ, Payne-Turner D, Tasian SK, Reshmi S, Cottrell CE, Reaman GH, Bowman WP, Carroll WL, Loh ML, Winick NJ, Hunger SP, Willman CL. Outcome modeling with CRLF2, IKZF1, JAK, and minimal residual disease in pediatric acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2012 Apr 12;119(15):3512-22. doi: 10.1182/blood-2011-11-394221. Epub 2012 Feb 24. PMID 22368272
- [Background] Rabin KR, Gramatges MM, Borowitz MJ, Palla SL, Shi X, Margolin JF, Zweidler-McKay PA. Absolute lymphocyte counts refine minimal residual disease-based risk stratification in childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2012 Sep;59(3):468-74. doi: 10.1002/pbc.23395. Epub 2011 Nov 18. PMID 22102553
- [Background] Xu H, Cheng C, Devidas M, Pei D, Fan Y, Yang W, Neale G, Scheet P, Burchard EG, Torgerson DG, Eng C, Dean M, Antillon F, Winick NJ, Martin PL, Willman CL, Camitta BM, Reaman GH, Carroll WL, Loh M, Evans WE, Pui CH, Hunger SP, Relling MV, Yang JJ. ARID5B genetic polymorphisms contribute to racial disparities in the incidence and treatment outcome of childhood acute lymphoblastic leukemia. J Clin Oncol. 2012 Mar 1;30(7):751-7. doi: 10.1200/JCO.2011.38.0345. Epub 2012 Jan 30. PMID 22291082
- [Background] Borowitz MJ, Devidas M, Hunger SP, et al.: Prognostic signficance of end consolidation minimal residual disease (MRD) in childhood acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG). [Abstract] J Clin Oncol 26 (Suppl 15): A-10000, 2008.
- [Background] Borowitz MJ, Devidas M, Hunger SP, Bowman WP, Carroll AJ, Carroll WL, Linda S, Martin PL, Pullen DJ, Viswanatha D, Willman CL, Winick N, Camitta BM; Children's Oncology Group. Clinical significance of minimal residual disease in childhood acute lymphoblastic leukemia and its relationship to other prognostic factors: a Children's Oncology Group study. Blood. 2008 Jun 15;111(12):5477-85. doi: 10.1182/blood-2008-01-132837. Epub 2008 Apr 3. PMID 18388178
- [Background] Davies SM, Borowitz MJ, Rosner GL, Ritz K, Devidas M, Winick N, Martin PL, Bowman P, Elliott J, Willman C, Das S, Cook EH, Relling MV. Pharmacogenetics of minimal residual disease response in children with B-precursor acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2008 Mar 15;111(6):2984-90. doi: 10.1182/blood-2007-09-114082. Epub 2008 Jan 8. PMID 18182569
- [Background] Hinds PS, Hockenberry MJ, Gattuso JS, Srivastava DK, Tong X, Jones H, West N, McCarthy KS, Sadeh A, Ash M, Fernandez C, Pui CH. Dexamethasone alters sleep and fatigue in pediatric patients with acute lymphoblastic leukemia. Cancer. 2007 Nov 15;110(10):2321-30. doi: 10.1002/cncr.23039. PMID 17926333
- [Background] Winick N, Martin PL, Devidas M, et al.: Delayed intensification (DI) enhances event-free survival (EFS) of children with B-precursor acute lymphoblastic leukemia (ALL) who received intensification therapy with six courses of intravenous methotrexate (MTX): POG 9904/9905: a Children's Oncology Group study (COG). [Abstract] Blood 110 (11): A-583, 2007.
- [Result] Chen I, Harvey R, Mullighan CG, et al.: Relationship of CRLF2 expression and outcome in pediatric B-cell precursor acute lymphoblastic leukemia (BCP-ALL): A report from the Children's Oncology Group. [Abstract] J Clin Oncol 29 (Suppl 15): A-9505, 2011.
- [Derived] Ramsey LB, Panetta JC, Smith C, Yang W, Fan Y, Winick NJ, Martin PL, Cheng C, Devidas M, Pui CH, Evans WE, Hunger SP, Loh M, Relling MV. Genome-wide study of methotrexate clearance replicates SLCO1B1. Blood. 2013 Feb 7;121(6):898-904. doi: 10.1182/blood-2012-08-452839. Epub 2012 Dec 11. PMID 23233662
- [Derived] Yang JJ, Cheng C, Devidas M, Cao X, Campana D, Yang W, Fan Y, Neale G, Cox N, Scheet P, Borowitz MJ, Winick NJ, Martin PL, Bowman WP, Camitta B, Reaman GH, Carroll WL, Willman CL, Hunger SP, Evans WE, Pui CH, Loh M, Relling MV. Genome-wide association study identifies germline polymorphisms associated with relapse of childhood acute lymphoblastic leukemia. Blood. 2012 Nov 15;120(20):4197-204. doi: 10.1182/blood-2012-07-440107. Epub 2012 Sep 24. PMID 23007406
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/